CLINICAL TRIAL: NCT07276048
Title: Community Genetic Navigation Engagement Specialists (CoGENES) Training Program
Brief Title: Community Genetic Navigation Engagement Specialists to Increase Knowledge About Colorectal Cancer Genetics in Hispanic/Latino/a Communities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 19PS-24-8; NCI-2025-02710 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19PS-24-8 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH); U2CCA252971-01A1 (NIH)
Record Dates: First submitted 2025-09-16; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Observational (Focus group) (Other): Participants attend a focus group, over 60-90 minutes, on study.
  Interventions: Other: Discussion
- Phase I (Education) (Experimental): Participants complete educational sessions regarding colorectal cancer genetics over 3 hours each, one to two times per week, for a total of 18 hours over 3-6 weeks. Participants may attend virtual check-in meetings over 30-60 minutes each month. Participants who complete the training program may then participate in phase II.
  Interventions: Other: Educational Intervention; Other: Interview; Other: Survey Administration
- Phase II (Training, education) (Experimental): Participants who completed phase I train additional participants via educational sessions regarding colorectal cancer genetics. New phase II participants attend the educational sessions regarding colorectal cancer genetics, led by phase I participants, over a total of 10-18 hours. Participants may attend virtual check-in meetings over 30-60 minutes each month.
  Interventions: Other: Educational Intervention; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Other: Discussion — Attend focus group
  Other Names: Discuss
  Arms: Observational (Focus group)
Other: Educational Intervention — Complete educational sessions
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Phase I (Education); Phase II (Training, education)
Other: Educational Intervention — Train participants
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Phase II (Training, education)
Other: Interview — Ancillary studies
  Arms: Phase I (Education); Phase II (Training, education)
Other: Survey Administration — Ancillary studies
  Arms: Phase I (Education); Phase II (Training, education)

SUMMARY:
This clinical trial tests how well an educational program for training Hispanic/Latino/a (H/L) community members regarding colorectal cancer genetics works to increase knowledge about genetic and genomic testing. H/L populations are underrepresented in colorectal cancer tumor and genetics studies due to lack of access of patients in clinical genetic testing, very low participation in clinical trials, lack of knowledge about cancer genetics and genomics, and lack of culturally sensitive materials for patient engagement in cancer genetics and genomic research. The community genetic navigation engagement specialist training program may increase knowledge regarding colorectal cancer genetics in H/L communities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate a genetic education program for H/L community health educators to train them as Community Genetic Navigation Engagement Specialists (CoGENES).

II. To evaluate a culturally tailored CoGENES Educational Tool Kit for H/L communities on genetic research, genetic counseling, and cancer risk assessments to be used by the CoGENES trainees to disseminate to community agencies.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of the CoGENES Educational program to improve the confidence of community health educators to train others in the community, as demonstrated by:

Ia. Self-confidence delivering training survey scores; Ib. Number of educators trained by each CoGENES; Ic. As well as the number of people reached in the community at large.

OUTLINE: Participants are assigned to 1 of 3 groups.

PHASE 1: Participants complete educational sessions regarding colorectal cancer genetics over 3 hours each, one to two times per week, for a total of 18 hours over 3-6 weeks. Participants may attend virtual check-in meetings over 30-60 minutes each month. Participants who complete the training program may then participate in phase II.

PHASE 2: Participants who completed phase I train additional participants via educational sessions regarding colorectal cancer genetics. New phase II participants attend the educational sessions regarding colorectal cancer genetics, led by phase I participants, over a total of 10-18 hours. Participants may attend virtual check-in meetings over 30-60 minutes each month.

FOCUS GROUP: Participants attend a focus group, over 60-90 minutes, on study.

After completion of study intervention, participants in phase I and II are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* SURVEYS (PHASE 1 AND 2) AND FOCUS GROUP: Must be 18 years of age or older
* SURVEYS (PHASE 1 AND 2) AND FOCUS GROUP: Ability to understand and the willingness to sign a written informed consent
* SURVEYS (PHASE 1 AND 2) AND FOCUS GROUP: Self-reported H/L ethnicity, of any race
* SURVEYS (PHASE 1 AND 2) AND FOCUS GROUP: Ability to read and write English or Spanish

Exclusion Criteria:

* SURVEYS (PHASE 1 AND 2) AND FOCUS GROUP: Any one younger than 18 years of age
* SURVEYS (PHASE 1 AND 2) AND FOCUS GROUP: Any person with major cognitive deficit or psychiatric impairment
* SURVEYS (PHASE 1 AND 2) AND FOCUS GROUP: Any person unable to read English or Spanish, and/or unable to write English or Spanish (for surveys participants only)
* SURVEYS AND FOCUS GROUP: No one younger than 18 years of age
* SURVEYS AND FOCUS GROUP: Any person with major cognitive deficit or psychiatric impairment
* SURVEYS AND FOCUS GROUP: Unable to read English or Spanish, and/or unable to write English or Spanish (for Surveys among CoGENES only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-12-11 (Estimated); Study Completion 2027-12-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants who completed training program | Up to 36 months
  Will report the number of participants started and number of participants who successfully completed the training program. Training is considered successful if they complete the required number of hours. Training lasts 3 hours per session once a week over 6 weeks. We will recruit 10-12 trainees per year for 3 years.
Knowledge gained after training | Up to 36 months
  After training, participants will be assessed about their knowledge of genetic testing before training new trainees and educating community members. Will use the Genetic Literacy and Comprehension (GLAC) measure to assess trainees knowledge with eight commonly used genetic terms and concepts (genetic, chromosome, susceptibility, mutation, variation, abnormality, heredity, and sporadic) using a 7-point scale of 1 "Strongly Disagree" to 7 "Strongly Agree". We will compare pre- and post- surveys to assess knowledge.
Confidence of training after training completion | Up to 36 months
  Measured by scores obtained from questioners developed by our team to capture confidence level of participants in training peers, focusing on confidence of explaining each module of the program to prospective trainees and answering questions, as well as confidence level using our Educational Toolkit to educate the community at large. Higher scores mean more confidence.
Number of people trained and/or reached in the community | At 6 and 12 month follow up
  Will report number of people trained and/or reached in the community
Completion of focus groups | Up to 2 years
  Will focus on readability, knowledge, acceptability, barriers. These qualitative analyses focus on the educational materials themselves, and their ability to transfer knowledge in the most effective way, as well as assessing the effectiveness of the materials in transferring information that is understandable, readable and usable for participants to train others.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Baezconde-Garbanati, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California